CLINICAL TRIAL: NCT00979719
Title: Improvement of a Physically Active Lifestyle in Orthopedic and Cardiologic Rehabilitation Patients With an Expert System
Brief Title: Improvement of a Physically Active Lifestyle
Acronym: FaBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Collaborators: Deutsche Rentenversicherung (Other)
Responsible Party: Sonia Lippke, Dr.; Assistant Professor (C1), Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 8011 - 106 - 31/31.91; 0421/00-40-64-50-00
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2011-01

CONDITIONS: Pain; Osteoarthritis; Rheumatoid Arthritis; Heart Diseases; Diabetes Mellitus, Type 2; Behavior; Motivation
Keywords: Randomized Controlled Trial; evidence- and theory-based behavioral intervention; expert system; stages of change; motivational interviewing; tailoring; Self Care; Rehabilitation; Expert Systems
MeSH Terms: conditions — Pain; Osteoarthritis; Arthritis, Rheumatoid; Heart Diseases; Diabetes Mellitus, Type 2; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention Group (IG) (Experimental): Patients in the IG will receive an interactive, computerized expert system which tailors treatment components to the individual needs of the patients
  Interventions: Behavioral: Intervention Group (IG)
- Active Control Group (ACG) (Placebo Comparator): Patients in the ACG will get an interactive computerized standard program which has been proven to be effective (Göhner, & Fuchs, 2007) Göhner, W. & Fuchs, R. (2007). Änderung des Gesundheitsverhaltens. MoVo-Gruppenprogramme für körperliche Aktivität und gesunde Ernährung. Göttingen: Hogrefe.
  Interventions: Behavioral: Active Control Group (ACG)
- Passive Control Group (PCG) (No Intervention): patients are asked to answer the questionnaires only

INTERVENTIONS:
Behavioral: Intervention Group (IG) — patients will receive an interactive, computerized expert system which tailors treatment components to the individual needs of the patients
  Other Names: FaBA
  Arms: Intervention Group (IG)
Behavioral: Active Control Group (ACG) — Patients in the ACG will get an interactive computerized standard program which has been proven to be effective (Göhner, W. & Fuchs, R. (2007). Änderung des Gesundheitsverhaltens. MoVo-Gruppenprogramme für körperliche Aktivität und gesunde Ernährung. Göttingen: Hogrefe.)
  Other Names: MoVo
  Arms: Active Control Group (ACG)

SUMMARY:
To help rehabilitation patients to adopt and maintain a physically active lifestyle, it is imperative to increase self-management competencies. Aim of this research project is to evaluate an evidence- and theory-based computerized expert system in comparison to a well established standard program and a questionnaire-only group. Rehabilitation patients will be treated psychologically and followed up over 18 months. The computerized expert system is expected to help patients better than the standard program. Both interventions are hypothesized to improve self-management competencies over and above the rehabilitation treatment (i.e., questionnaire-only group).

DETAILED DESCRIPTION:
An experimental study with three groups is planned over a time period of 18 months. Patients in the intervention group receive an interactive, computerized expert system (Intervention Group, IG). Patients in the Active Control Group (ACG) get an interactive computerized standard program. This standard program has already been proven to be effective but which does not tailor treatment components to the individual needs of the patients. Patients in the Passive Control Group (PCG) are asked to answer the questionnaires only. Rehabilitation patients (N = 1000) will be recruited in three rehabilitation clinics and followed up over six measurement points: t1 and t2 with computer interventions during their rehabilitation stay; t3 and t4 with booster-sessions via telephone (6 weeks and 6 months after admission from rehabilitation). Furthermore, patients will be contacted at t5 per mail with motivational material (12 months after admission) and at t6 again per mail (only questionnaire, 18 months after admission).

The hypotheses are: In comparison to the PCG, both the IG and the ACG are expected to have a higher motivation, to adopt a healthy lifestyle, to perform more health behavior and to be less likely to relapse into previous unhealthy routines. Also, IG and ACG will be healthier as well as they will report more quality of life and rehabilitation satisfaction. In comparison to ACG, the IG is hypothesized to be more effective than the ACG regarding motivation, behavior and social-cognitive predictors of behavior. Moreover, the interventions (ACG and IG) are supposed to be equally effective for cardiac and orthopedic, as well as out-patient and stationary treated rehabilitation patients. After successful evaluation and some adoptions the intervention will be implemented as a self-help program in all eligible rehabilitation clinics and in the internet.

ELIGIBILITY:
Inclusion Criteria:

* to be capable of exercising on their own at the minimum level recommended by the according rehabilitation clinic
* able to fill out a questionnaire (no illiteracy)
* adequate German language ability

Exclusion Criteria:

* the participant not be of age
* severe cognitive deficits
* visual impairments (patients have to read at the PC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1377 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
physical activity | 18 months

SECONDARY OUTCOMES:
subjective health | 18 months
quality of life | 18 months
rehabilitation satisfaction | 18 months
motivation | 18 months
social-cognitive predictors of behavior (self-efficacy, action control etc.) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, PhD, Principal Investigator — Freie Universitaet Berlin
Locations (1):
- Freie Universitaet Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Lippke S, Pomp S, Fleig L. Rehabilitants' conscientiousness as a moderator of the intention-planning-behavior chain. Rehabil Psychol. 2018 Aug;63(3):460-467. doi: 10.1037/rep0000210. PMID 30113201
- [Derived] Fleig L, Kerschreiter R, Schwarzer R, Pomp S, Lippke S. 'Sticking to a healthy diet is easier for me when I exercise regularly': cognitive transfer between physical exercise and healthy nutrition. Psychol Health. 2014;29(12):1361-72. doi: 10.1080/08870446.2014.930146. Epub 2014 Jul 21. PMID 24894668
- [Derived] Fleig L, Lippke S, Pomp S, Schwarzer R. Intervention effects of exercise self-regulation on physical exercise and eating fruits and vegetables: a longitudinal study in orthopedic and cardiac rehabilitation. Prev Med. 2011 Sep;53(3):182-7. doi: 10.1016/j.ypmed.2011.06.019. Epub 2011 Jul 14. PMID 21784096